CLINICAL TRIAL: NCT04367870
Title: COVID-19 Serodiagnosis in Oncology
Brief Title: COVID-19 Detection Test in Oncology
Acronym: EVIDENCE
Status: Completed | Type: Observational
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Other Study IDs: UC-TRA-2002; 2020-A01002-37 (Other: ID RCB)
Record Dates: First submitted 2020-04-28; First posted 2020-04-29 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Oncology
Keywords: Cancer; SARS-CoV-2; COVID-19; coronavirus; serodiagnosis; immunoassay
MeSH Terms: conditions — Neoplasms; COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non immune patient: Patients with a negative SARS-CoV-2 immunoassay
- Immune patient: Patients with a positive SARS-CoV-2 immunoassay

SUMMARY:
EVIDENCE is a non interventional, French, multicenter study. Patients will be screened by local severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) immunoassay in their oncology department (rapid diagnostic test (RDT) or enzyme-linked immunosorbent assay (ELISA)). In patients with positive local SARS-CoV-2 immunoassay, a centralized SARS-CoV-2 ELISA will be performed in order to double check the immune response of all patients considered immune by local immunoassay.

DETAILED DESCRIPTION:
Patients with cancer are a high-risk group in the COVID-19 pandemic. They are already vulnerable to infection because of their underlying illness and often immunosuppressed status, and are at increased risk of developing severe complications from the virus, including intensive care unit admission or even death. In light of this increased risk, many guidelines have been issued, aiming at minimizing the risk of SARS-CoV-2 infection occurrence and/or gravity. These changes in cancer care could however translate in less efficient or delayed treatments. In this study, we want to detect cancer patients that were exposed to the SARS-CoV-2 virus and acquired an immunity. These patients immune to the SARS-CoV-2 virus are susceptible to receive the standard of care, meaning the most appropriate treatment to manage their cancer. Large-scale serodiagnosis are considered as the solution to progressively relax the current lockdown in France. RDT and ELISA, which were not available until mid-April 2020, will be largely used in the general French population over the coming months, millions of tests have already been ordered by French authorities and companies.

The aim of this study is to control that oncology patients qualified immune by local immunoassay are indeed safe (i.e. have extremely low risk of SARS-CoV-2 infection following a positive local immunoassay test). Of note, several immunoassays (RDT or ELISA) will be used in the participating centers throughout the study. A confirmation of positive cases yielded by these different immunoassays will be performed by a centralized ELISA, in order to minimize the risk of false positive results.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years old
2. Patient diagnosed with invasive cancer (solid tumor only)
3. Patient in active phase of cancer treatment (surgery, chemotherapy, radiotherapy, immunotherapy or targeted therapy ongoing or planned within the next month- excepted patient treated by hormonotherapy and targeted therapy alone in adjuvant setting)
4. Patient with a local immunoassay realized before inclusion realized during the standard practice with a positive or negative result (test name and reference should be available)
5. Information and non-opposition of the patient to the study procedure

Exclusion Criteria:

1. Person deprived of their liberty or under protective custody or guardianship
2. Patients unwilling or unable to comply with the medical follow-up required by the study because of geographic, familial, social, or psychological reasons
3. Patients treated for a hematological malignancy
4. Life expectancy <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of individuals aged 18 years or older, in an active phase of treatment for any invasive cancer.
Sampling Method: Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2020-05-23 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the ability of SARS-CoV-2 immunoassays, following a positive result, to identify patients with very low risk of recurrence of COVID-19 within 3 months. | 3 months
  The primary endpoint of this study is the recurrence of COVID-19 within 3 months following the immunoassay-positive result obtained before the inclusion in the study. The recurrence is defined by the presence of symptoms confirmed either by a positive reverse transcription-polymerase chain reaction (RT-PCR) result for SARS-CoV-2 or by the adjudication committee. Immunoassay will be said positive as per the predefined reference corresponding to the immunoassay.

SECONDARY OUTCOMES:
To estimate the discordance rate between local immunoassay and a centralized ELISA in patients with a positive immunoassay, whatever the immunoassay. | 6 months
  Agreement between the different immunoassays and the centralized ELISA, using the centralized ELISA as benchmark.
To identify patients with very low risk of recurrence of COVID-19 within 6 months following a positive immunoassay result. | 6 months
  COVID-19 recurrence within 6 months following an immunoassay-positive result.
To characterize the evolution over time of the serologic response against SARS-CoV-2 (in a subgroup of patients). | 6 months
  Quantitative and qualitative detection of SARS-CoV-2-related antibodies and immune serum markers at baseline, 2-3 months and 4-6 months post-inclusion, in a subgroup of 200 patients.

CONTACTS AND LOCATIONS:
Overall Officials: François-Clément BIDARD, Principal Investigator — Institut Curie
Locations (7):
- France (7):
  - Centre Hospitalier de Boulogne sur Mer, Boulogne-sur-Mer
  - Centre Jean Perrin, Clermont-Ferrand
  - Hopitaux Civils de Colmar, Colmar
  - Hôpital Universitaire Pitié Salpêtrière, Paris
  - Institut Curie, Paris
  - Centre Eugène Marquis, Rennes
  - Institut Curie, Saint-Cloud

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.